Title: Researching Resiliency in Stressful Experiences (RISE) Program for Men Leaving Incarceration

NCT #: NCT04785677

Date: 5/17/2021

### Permission to Take Part in a Human Research Study



## Permission to Take Part in a Human Research Study

**Title of research study:** Researching the RISE Program for Men Leaving Incarceration

Investigator: Carrie Davis, PhD

**Key Information:** This is a summary of the study. It will help you chose if you want to be a part of this study. More detailed information is listed later on in this form.

### Why am I being invited to take part a research study?

We invite you to participate in this research study because you are a male between the ages of 18 and 35, will be released from a Florida Department of Corrections facility, and anticipate releasing to Columbia, Duval, Leon, or Suwanee county.

This study is not being conducted by Florida Department of Corrections (FDC). Corrections, law enforcement or the court will not get a copy of your name or of your answers. This study is being conducted by a research team at Florida State University.

#### What should I know about a research study?

Please review this consent information carefully. We provide information about the study that you should think about before deciding whether to take part. We include special information about steps that we will take to prevent your exposure to Coronavirus (COVID-19) when you take part in our face-to-face study activities.

- Someone will explain this research study to you.
- The study uses random assignment (sort of like using a toss of a coin) to either put you in the Resilience in Stressful Experiences (RISE) or a Reentry Services as Usual Group (RSU).
- If you do or do not take part is up to you.
- You can choose not to take part.
- You can choose to take part and later change your mind.
- Your decision will not be held against you.
- You can ask all the questions you want before you decide.
- Sentence length or supervision status will not be affected regardless of whether you choose to participate or not.
- This study is funded by the National Institute of Justice.

### Why is this research being done?

The study is to see if a program that starts in prison and keeps going after release from prison helps young men age 18-35 who have experienced extremely stressful life events after they are released from prison. We are testing a program called Resilience in Stressful Experiences (RISE) to see if it helps with some things that you may or may not have experienced such as: difficulties with stable employment or housing, impulsivity, aggression, coping, mental health, substance abuse and lowering the chance of returning to prison.

# Permission to Take Part in a Human Research Study How long will the research last and what will I need to do?

You will likely be participating in this study for up to 18 months.

Before you sign the consent form we will tell you about two different services: RISE and the usual reentry services that you would typically receive. You will be asked questions to see if you are able to take part in the study. If you are eligible to be in the study, you will either be in the RISE Group or the RSU Group. We will answer any questions you have about the RISE services. If you are in the RSU Group, we will still meet with you for follow-up interviews. However, you will not attend the same meetings that the RISE group attends. More detailed information about the study procedures can be found under "what happens if I say yes, I want to be in this research?"

### Is there any way being in this study could be bad for me?

You might experience distress related to the questions we ask you about your health, mental health or substance use. You do not have to talk about personal information if you choose not to.

In addition, there may be risks by having you take part in our face-to-face study activities during this time of Coronavirus. We have an information sheet describing the ways that we are reducing these risks for all involved with this study.

More information about the risks of participating in this study can be found under "Is there any way being in this study could be bad for me? (Detailed Risks)"

### Will being in this study help me in any way?

There are no certain benefits to you or others from being in this research. You may benefit from the program that this study is researching. If you are in the RISE group, you may benefit from its services. Or you may benefit from RSU which is the standard reentry services provided by FDC.

Being in this research study will not improve your housing or job while in prison. Being in this study will not affect any conditions to community supervision, if that applies. Being in this study will not affect your release date.

### What happens if I do not want to be in this research?

You can choose to be in or not be in the study. If you do not want to be in the study, you will be able to get any services regularly offered to people getting out of prison.

# **Detailed Information:** The following is more information about this study.

### Who can I talk to?

If you have questions, concerns, or complaints, or think the research has hurt you, talk to the research team at 850-645-2829 or by email at cpettusdavis@fsu.edu. The principle researcher's office is at Florida State University, Institute for Justice Research and Development, Tallahassee, FL 32310.

This research has been reviewed and approved by an Institutional Review Board ("IRB"). You may talk to them at 850-644-7900 or humansubjects@fsu.edu if:

- Your questions, concerns, or complaints are not being answered by the research team.
- You cannot reach the research team.
- You want to talk to someone besides the research team.
- You have questions about your rights as a research subject.
- You want to get information or talk about this research.

# Permission to Take Part in a Human Research Study How many people will be studied?

We will have 400 people to be in the research study, 200 in the RISE Group and 200 in the RSU Group with standard re-entry supports from Corrections and the community to which they are released.

## What happens if I say "yes" to being in this research?

First, we will talk with you about the study. You can ask any questions you have about the study.

Second, we ask you to sign this consent form.

Third, we will ask questions about past events in your life such as your education and work experiences, social life experiences, relationships with others, mental health and substance use experiences, and how you handle stress or other characteristics you perceive about yourself. A member of the research team will read to you from interview forms using a tablet. You will likely spend about an hour or two answering these questions and a contact form, which will help us in reaching you after you have gotten out of prison. The contact form includes asking about relatives and other persons who may be helpful in locating you for follow-up interviews.

Fourth, in the personal data we collect from you, we will replace your FDC identification number with a random meaningless number. This research number will help us to protect your personal identity and will allow us to keep track of your progress. This will help us see if being in RISE or RSU helps people. We will collect your name, birthdate, and correctional facility identification number. Everything you tell the researchers will be highly confidential.

Fifth, after you finish this first interview you will be randomly assigned either to the RISE Group or to the RSU Group. The group you get will be by chance, like flipping a coin. Neither you nor the researchers will choose what group you get. You will have an equal chance of being given in either group. We won't use your interview answers to affect which group you are in.

Sixth, if assigned to the RISE Group, you will be in the RISE program for up to 4 meetings while in prison, and up to 15 meetings after getting out of prison. If assigned to the RSU group you will receive the usual re-entry supports offered by Corrections or the community to which you are released.

Regardless of which group you are randomly assigned, you will be interviewed three times after you release from prison. We will ask you questions within the first two weeks of your release and then again, and then approximately four months later, and then again four months after that (approximately 8 months after release from prison).

Throughout the study, we will get information from the FDC and other government databases about you. This will include information about your: date of birth, race/ethnicity, marital status, level of education, age at first offense, number of previous incarcerations, most serious offense, program and treatment participation while incarcerated or during supervision, infractions, and current sentence length. Additionally, we will receive expected release data, primary language, county of conviction, most recent admission date, Spectrum assessment date, and Spectrum risk index score from the FDC as a part of the recruitment process. We will also get your social security number from FDC. The reason for getting your social security number is to be able to keep track of you while in and after getting out of prison. Social security numbers are better at tracking records than only relying on birthdate. All of these personal identifiers are retained separate from the research data until data analysis but your personal identifiers will not be revealed to anyone beyond the research team or in any analysis.

# Permission to Take Part in a Human Research Study What happens if I say "yes, but I change my mind later?

You can leave the study at any time and it will not be held against you.

### Is there any way being in this study could be bad for me? (Detailed Risks)

If you are in the RISE program, talking about your past may bring up emotions and may be uncomfortable. You may have a lot of feelings when thinking about past life events. If you feel you need help with these feelings, please let a team member know. While still in prison, you should let your classification staff member know you need mental health services. Once you are released, we have provided resources at the end of this consent form that may assist you in finding mental health services for research-related distress.

One risk is that information about you may be revealed by mistake. We will use our best efforts to keep information about you private. We do not work for the Florida Department of Corrections, and nothing that can identify you that we collect will be shared with Florida Department Corrections employees. The research team will keep private the information you give. Answers you give and what you talk about in this study are private. But, if you talk about hurting yourself, hurting somebody else, escaping from prison, or in-prison sexual assault we may have to share this information with professionals either to comply with the law or to get you to services you might need.

While we do not directly ask about in-prison sexual contact, all study team members are trained in the Prison Rape Elimination Act (PREA), which the team has to do to be given access to the prisons. All PREA rules for the facility will be followed at all times.

When you get out of prison, if you are feeling suicidal or think you are going through a crisis and want some help from a professional, please call the national suicide hotline at 1-800-SUICIDE or 1-800-272-TALK.

There may be risks that we do not know about. You should tell any problems you may have to the researcher.

# What happens to the information collected for the research?

We will do everything we can to not reveal your personal information to people who have a need to see this information. Groups that may look at your information include the IRB and other members of this organization.

Your name will not be in surveys, only a meaningless research code number. These surveys will be kept securely in a data storage system called REDCap. Additionally, de-identified study data will be archived at the National Archive of Criminal Justice Data (NACJD). Only the research team members and the Principal Investigator can get the code number.

A member of the research team will obtain a list of names of possible participants from FDC. A secure location at the prison will be used for the interviews to make sure we guard your privacy. The RISE Group meetings will also be private and confidential.

Prison staff are not a part of this project. They will not get a copy of your name or of your answers.

### Permission to Take Part in a Human Research Study

Prison administrators will receive a copy of the results at the end of the study but will not be able to identify you personally from what they get.

#### This research is covered by a DOJ Privacy Certificate from the National Institute of Justice.

This means that we cannot release or use information, documents, or samples that may identify you in any action or lawsuit unless you give permission to do this in writing. This protection means that no court can order your information to be released to the court or any other party. This protection includes federal, state, or local civil, criminal, administrative, legislative, or other legal proceedings.

### Can I be removed from the research without my OK?

Your signature documents your permission to take part in this research.

You can be removed from the research study without your say. Reasons for removal include preventing research from being carried out or no longer meeting requirements.

We will tell you about any new information that may affect your health, welfare, or choice to stay in the research.

#### What else do I need to know?

You will not get anything for taking part in this study while in prison. You will get \$25 dollars each time you finish the post-release interviews for a total of \$75. Additionally, if you are in the RISE group you will have the opportunity to receive up to \$10.00 gift card for every RISE session you complete with research staff post incarceration. The amount of the gift card will be selected by lottery. There will be three \$10.00 gift cards and two \$5.00 gift cards for every five participants. You will not get money for completing RISE program sessions while incarcerated.

| Signature of subject | Date |
|---|---|
| Printed name of subject | _ |
| Signature of person obtaining consent | Date |
| Printed name of person obtaining consent | _ |
| | 1:1 (21 2:12 1 |
| Your signature documents you acknowledge the circumstances unde<br>broken. Certain situations described in this consent may mean the stunformation about you. If you share information about being sexual a | ady will need to release some |
| | cidal intent or intent to cause |

# Signature of subject Date Printed name of subject Signature of person obtaining consent Date Printed name of person obtaining consent Your signature documents your permission to take part in this research. Signature of subject Date Printed name of subject Signature of person obtaining consent Date Printed name of person obtaining consent Your signature documents you acknowledge the circumstances under which confidentiality can be broken. Signature of subject Date Printed name of subject Signature of person obtaining consent Date Printed name of person obtaining consent

Permission to Take Part in a Human Research Study